CLINICAL TRIAL: NCT07312656
Title: Aerosolized Mesenchymal Stem Cell-Derived Exosomes for the Prevention and Treatment of Radiation-Induced Oral Mucositis: A Randomized Controlled Trial
Brief Title: Aerosolized Mesenchymal Stem Cell-Derived Exosomes for the Prevention and Treatment of Radiation-Induced Oral Mucositis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Guangxi Medical University (Other)
Collaborators: LiuZhou People's Hospital (Other); First People's Hospital of Yulin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-K0439
Record Dates: First submitted 2025-12-05; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Oral Mucositis (Ulcerative) Due to Radiation
MeSH Terms: conditions — Stomatitis; Ulcer

STUDY DESIGN:
Intervention Model Description: The stratified block randomization method was employed to ensure balanced baseline characteristics between groups and the unpredictability of random allocation.
Masking Description: This study adopted an open-label design, meaning that both the investigators and the participants are aware of the treatment group assignments. The investigational and control medications were not processed for blinding purposes and were routinely provided and used in their standard forms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): mesenchymal stem cell-derived exosomes. Administer the mesenchymal exosome spray three times daily-30 minutes after each main meal (breakfast, lunch, and dinner)-with a dosage of approximately 1.5 mL per application. Initiation of the study drug on the first day of radiotherapy and continuing through the completion of the treatment course.
  Interventions: Drug: mesenchymal stem cell-derived exosomes
- control group (No Intervention): Patients in the control group received no drug interventions, only conventional radiotherapy and supportive care.

INTERVENTIONS:
Drug: mesenchymal stem cell-derived exosomes — Mesenchymal Exosome Administration Protocol: 1. Administration Timing: Begin 7 days prior to radiotherapy initiation and continue until 14 days post-radiotherapy completion. 2. Preparation: Remove the exosome vial, open the cap, add 5mL of saline solution, and secure the spray cap. 3. Administration Frequency: 3 times daily (30 minutes after breakfast, lunch, and dinner). 4. Dosage: Approximately 1.5mL per spray. 5. Administration Method: Oral spray. Evenly spray onto the oral mucosal surface. Avoid eating or rinsing for 20 minutes after administration.
  Arms: experimental group

SUMMARY:
Radiation-induced oral mucositis (RIOM) is an inevitable acute complication in radiotherapy for head and neck malignancies, characterized by a complex pathogenesis involving multiple biological processes. According to the latest data from the International Agency for Research on Cancer (IARC), approximately 650,000 new cases of head and neck cancers are diagnosed globally each year, with about 70% of patients undergoing radiotherapy. RIOM develops through a multistep pathophysiological cascade, including initiation of mucosal injury, signaling amplification, inflammatory response, ulceration, and eventual healing. Ionizing radiation induces DNA damage in oral mucosal epithelial cells, triggering increased apoptosis. This cellular injury promotes the activation and release of pro-inflammatory mediators such as tumor necrosis factor-α (TNF-α), interleukin-1β (IL-1β), and interleukin-6 (IL-6), compromising the integrity of the mucosal barrier and ultimately leading to ulcer formation. Current clinical management of RIOM remains largely supportive, relying on oral hygiene, nutritional supplementation, and pain control, with no effective prophylactic agents available. Despite extensive research into potential interventions internationally, no drugs specifically approved by the FDA or NMPA for the prevention of RIOM have reached the market. This significant unmet clinical need calls for urgent scientific and therapeutic advancement. This study aims to evaluate the therapeutic efficacy and safety profile of aerosolized exosomes derived from mesenchymal stem cells in the prevention and treatment of radiation-induced oral mucositis in patients receiving radiotherapy for head and neck cancers. The ultimate objective is to establish a novel and effective therapeutic strategy for clinical application.

DETAILED DESCRIPTION:
This study employs a randomized controlled design, aiming to enroll a total of 200 head and neck cancer patients scheduled to undergo radiotherapy from three medical centers. The experimental group (100 patients) will receive a mesenchymal stem cell-derived exosome spray, while the control group (100 patients) will follow a placebo-controlled design without any pharmacological intervention, receiving only standard radiotherapy and supportive care. The primary endpoint is the incidence of grade 3 or higher radiation-induced oral mucositis, which will be used to evaluate the efficacy of the investigational agent in preventing and ameliorating this condition through comparison with the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed malignant tumor of the head and neck;
2. Age 18-75 years;
3. Scheduled to receive radical radiotherapy with a total planned dose of ≥60 Gy, with radiation fields including the oral cavity and/or oropharynx;
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2 and a life expectancy of ≥6 months.
5. White blood cell≥3.0×10^9/L, hemoglobin≥ 90 g/L, platelet (PLT)≥ 100x10^9/ L
6. Transaminases≤2.5 times the upper limit of normal, total bilirubin ≤1.5 times the upper limit of normal;
7. Serum creatinine ≤1.5 × ULN or creatinine clearance ≥50 mL/min;
8. Cardiac: Electrocardiogram (ECG) without clinically significant abnormalities;
9. Intact oral mucosa before initiation of radiotherapy. Absence of active oral infections or severe periodontal disease before initiation of radiotherapy;
10. Signed informed consent form.

Exclusion Criteria:

1. Previous radiotherapy to the head and neck region;
2. Head and neck surgery within the preceding 4 weeks;
3. Current participation in another clinical trial, or participation in another interventional study within the past 4 weeks;
4. Significant cardiovascular disease, including unstable angina, myocardial infarction within the past 6 months, severe arrhythmia, or heart failure (NYHA Class III-IV);
5. Severe hepatic or renal dysfunction, such as cirrhosis or chronic renal insufficiency (creatinine clearance <30 mL/min);
6. Active systemic infection requiring antimicrobial therapy;
7. Autoimmune diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis) requiring ongoing immunosuppressive treatment;
8. Severe psychiatric disorders that may impair the ability to provide informed consent or adhere to the study protocol;
9. Using other oral mucosal protective agents or anti-inflammatory medications that cannot be discontinued. Long-term use of immunosuppressants or corticosteroids at a prednisone-equivalent dose >10 mg/day;
10. Individuals unable to comprehend the study requirements or comply with study procedures;
11. Any other condition that, in the judgment of the investigator, would render the patient unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade ≥3 radiation-induced oral mucositis | Within 90 days from the initiation to the completion of radiotherapy
  The primary endpoint is defined as the proportion of patients who develop grade 3 or higher radiation-induced oral mucositis (RIOM) from the start of radiotherapy until 90 days after the completion of radiotherapy. RIOM was graded according to the WHO oral toxicity scale criteria: Grade 0: No changes in the oral mucosa; Grade 1: Erythema of the oral mucosa with mild pain, not requiring analgesics; Grade 2: Patchy mucositis with serous exudate, moderate pain, usually not requiring analgesics; Grade 3: Confluent mucositis with severe pain requiring analgesics; Grade 4: Ulceration, hemorrhage, or necrosis, with intense pain affecting oral intake.

SECONDARY OUTCOMES:
Incidence rate of RIOM at any level | Within 90 days from the initiation to the completion of radiotherapy
  Assess the difference in the proportion of patients experiencing any grade (Grade 1 or higher) of RIOM between the intervention group and the control group to evaluate the overall preventive efficacy of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China